CLINICAL TRIAL: NCT05285878
Title: A Phase 2, Randomized, Placebo-Controlled Study to Evaluate Fingolimod for the Abrogation of Interstitial Fibrosis and Tubular Atrophy Following Kidney Transplantation
Brief Title: Fingolimod for the Abrogation of Interstitial Fibrosis and Tubular Atrophy Following Kidney Transplantation
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Ahmed Osama Gaber, MD, Chair, Department of Surgery, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO00022269; U1111-1226-4680 (Registry Identifier: World Health Organization)
Record Dates: First submitted 2022-03-08; First posted 2022-03-18 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Interstitial Fibrosis; Kidney Transplant; Complications; Kidney Transplant Rejection; Kidney Transplant Failure and Rejection; Kidney Transplant Failure; Kidney Failure, Chronic; Graft Rejection
Keywords: Fingolimod Hydrochloride; Kidney Transplantation; Glomerular Filtration Rate; Kidney; Fibrosis; Immunosuppression Therapy; TOR Serine-Threonine Kinases; Graft Survival; Transplantation; Transplant Recipients; Organ Transplant; Tubular Atrophy; Interstitial Fibrosis and Tubular Atrophy
MeSH Terms: conditions — Pulmonary Fibrosis; Rejection, Psychology; Kidney Failure, Chronic; Fibrosis | interventions — Fingolimod Hydrochloride; Methylcellulose

STUDY DESIGN:
Intervention Model Description: Phase 2, Randomized, Placebo-Controlled Study
Who Masked: Participant, Care Provider
Masking Description: Participants and the study team will be blinded as to the assignment until the database is locked. Only the investigational pharmacist will know the study assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants will take a placebo capsule daily for 3 months. Placebo will be methylcellulose encapsulated into an opaque closed gelatin capsule for blinding. Capsules will be placed in a labeled bottle, with the contents only identifiable by a code on the package label and only the compounding pharmacy and the unblinded pharmacist at Houston Methodist Investigational Drug Service will know the code definition.
  Interventions: Drug: Placebo
- Fingolimod (Active Comparator): Participants will take a 0.5 mg fingolimod capsule each day for 3 months. The fingolimod capsule will be placed inside an opaque closed gelatin capsule without transformation of the manufacteror's fingolimod capsule. The fingolimod blinded product and the placebo capsule will be identical in size, color, appearance, and weight.
  Interventions: Drug: Fingolimod

INTERVENTIONS:
Drug: Fingolimod — 0.5 mg daily
  Other Names: GILENYA®; FTY720
  Arms: Fingolimod
Drug: Placebo — 0.5 mg daily
  Other Names: methylcellulose
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled trial in de novo kidney transplant patients to determine if the addition of fingolimod (brand name Gilenya®, candidate name- FTY720) on the background of standard immunosuppression will prevent expansion of the interstitial compartment of the transplanted kidney. Interstitial expansion is the precursor of interstitial fibrosis and graft loss. The study will test the hypothesis that abgrogating the fibrogenic effects of both the RhoA and mTOR pathways with fingolimod will reduce structural damage in transplanted kidneys and possible subsequent transplant failure.

DETAILED DESCRIPTION:
Prevention of, or slowing the progression of, the development of allograft fibrosis has not been successful in previous efforts. This study will to evaluate the potential of fingolimod (Gilenya®, Novartis Pharmaceuticals, East Hanover, NJ) (1), a sphingosine 1-phosphate receptor modulator and a RhoA inhibitor (2), to abrogate the presence of interstitial fibrosis/tubular atrophy (IF/TA) after kidney transplantation. The study may provide important information for future clinical trials for prevention of IF/TA in kidney transplant recipients.

Interstitial fibrosis and tubular atrophy almost invariably occur together (10) and are present in approximately 45% of kidney allografts by the first year posttransplant (11). Naesens et al (11) demonstrated that any positive chronic interstitial fibrosis score is associated with graft loss after the first year post transplant with a more rapidly declining slope than those without interstitial fibrosis. Furthermore, they demonstrated that a tubular atrophy score of 2-3 was associated with 20% graft loss during the 2nd year posttransplant, >30% graft loss by 5 years and ~60% graft loss by 10 years posttransplant. Combined, IF/TA contributes to renal graft dysfunction or the decline in kidney function after transplantation and may be a factor in the 20.6% of total grafts lost (including death) by 5 years post-transplant (11,12).

Expansion of the interstitial compartment is a major component of IF/TA. Protocol (12,13) and for-cause (10,11) biopsies have provided evidence of the worsening of IF/TA with time in kidney transplant recipients and demonstrated a direct relationship between interstitial expansion and renal allograft functional decline and graft failure (11-14). Assessing the interstitial expansion by quantifying the fraction of renal cortical volume:interstitial compartment changes over time standardizes the assessment of IF/TA (15,16) and will be used in the current protocol (Section 10.2.1).

Fingolimod was originally intended as a prophylaxis against acute rejection in transplant recipients (17). A full development program was produced beginning with pharmacokinetics of single dose (18) and multiple doses (19) in healthy volunteers and evaluations of the effect of FTY720 on T-lymphocytes to better understand the immunosuppressive properties of the sphingosine 1-phosphate receptor modulator (20). Development proceeded with several studies where fingolimod was compared to standard immunosuppression regimens as an adjunct therapy with calcineurin inhibitors for prevention of kidney transplant acute rejection. After two cardiac events occurred in an open-label trial and lack of efficacy for prevention of acute rejection was demonstrated, the development of fingolimod as a therapeutic agent for rejection prophylaxis in transplantation ceased. Whereas the current study is not proposed to prevent acute rejection and will be using a smaller dose than those evaluated in phase 3 trials for acute rejection prophylaxis, a summary of these studies is important to the understanding of the safety of fingolimod in kidney transplant recipients.

Studies of de novo kidney transplant recipients report a reduction in absolute lymphocyte counts of approximately 25-35% in the lower dose groups (0.25mg and 0.5mg FTY720, respectively) that corrects to within approximately 20% of baseline (day of transplant surgery) level (22-28). Additionally, asymptomatic bradycardia or reduced heart rate was reported and responded to treatment when required or resolved on its own (23-26,28). Prudent exclusion criteria of patients who have heart rate <50bpm at baseline is warranted for the current study. Macular edema occurred more often in kidney transplant patients taking ≥2.5mg FTY720 (15/667, 2.2%) compared to mycophenolate mofetil (MMF, 5/373, 1.3%; 25,26,28); thus, the current study will exclude patients with a history of macular degeneration or diabetic retinopathy. Only one report indicated that liver enzymes were elevated in participants taking FTY720 (25) and the increase was mild (<2x upper limit of normal [ULN]).

Controlling hypertension and prevention and treatment of acute rejection are standard approaches to kidney function preservation in kidney transplant recipients. Additionally, the use of calcineurin inhibitor (CNI)-sparing protocols has been reported with various approaches but data are insufficient to equivocally demonstrate consistently lower IF/TA in the approaches reported to date (7). Thus, it is important to examine additional approaches for prevention of IF/TA in this population.

Preliminary data from Chen W et al strongly suggests that fingolimod is able to inhibit chronic rejection of transplanted hearts in a rat and mouse model by inhibiting RhoA and down-regulating mammalian target of rapamycin (mTOR) Complex 2 (mTORC2)/Regulatory Associated Protein Of MTOR Complex 1 Independent Companion Of MTOR Complex 2 (RICTOR; 30,31). Therefore, this study will test the hypothesis that abrogating the fibrogenic effects of both RhoA and mTOR pathways with fingolimod would abrogate IF/TA and that reducing this structural damage in transplanted kidneys would result in improved or preserved kidney function and reduced graft loss.

The purpose of this study is to demonstrate that 0.5mg/day of fingolimod for 3 months administered to de novo kidney transplant recipients will be safe and to examine the course of IF/TA over a 1-year period by testing the ability of 0.5mg/day fingolimod for 3 months to abrogate the development of IF/TA in de novo kidney transplant recipients compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Receiving a first or second kidney transplant
* Male or female, aged ≥18 to ≤65
* Women of child bearing potential who have a negative serum pregnancy test prior to treatment
* Women of child bearing potential (including perimenopausal women who have had a menstrual period within the previous 1 year) who agree to use 2 forms of effective birth control regimen (at least one of which is a barrier method) throughout the study period and for 6 weeks following the end of the study or the last dose of mycophenolic acid, whichever comes first.
* Panel of reactive antibodies <50%
* Able to take oral medication
* Agreement to adhere to Lifestyle Considerations throughout study duration: refraining from the consumption of grapefruit or grapefruit juice and stopping any anticoagulation therapy, including ASA, one week prior and one week post kidney biopsy procedure

Exclusion Criteria:

* Transplantation of any organ other than kidney
* History or presence of second degree AV block, third degree AV block, symptomatic bradycardia, or an arrhythmia requiring current treatment with Class Ia or III antiarrhythmic drugs.
* Heart rate <60 beats per minute
* Presence of an increased QTc interval > 500 ms on screening ECG.
* Presence of a cardiac pacemaker.
* History of any major cardiac events, including heart attack within the last six months of enrollment, unstable angina, congestive heart failure, or any severe cardiac disease as determined by investigator
* Known macular degeneration
* Diagnosed with any significant coagulopathy or medical condition requiring long-term systemic anticoagulation after transplantation, which would interfere with obtaining biopies.
* Diagnosed with chronic immune system disease
* Diagnosed with acute pulmonary disease
* Diagnosed with severe liver disease, including abnormal liver enzymes or total bilirubin greater than three times upper limit of normal.
* Diagnosed with any past or present malignancies except squamous or basal cell carcinoma of the skin excised at least two years prior to randomization.
* Diagnosed with active acute or chronic infection, or febrile illness within two weeks prior to randomization.
* Recent history of strokes in the preceding 6 months
* Use of ketoconazole for more than 2 weeks
* Use of any investigational drug during the 4 weeks prior to enrolling in this study
* Women of child bearing potential who are breastfeeding
* Women of childbearing potential not practicing reliable methods of contraception. Reliable methods for contraception include surgical sterilization (hysterectomy, bilateral tubal ligation), double-barrier method (such as condom and diaphragm). To be considered as post-menopausal and not of childbearing potential, female participants must have experienced 12 consecutive months of amenorrhea.
* Known allergic reactions to components of Gilenya®, specifically fingolimod, gelatin, magnesium stearate, mannitol, titanium dioxide, and/or yellow iron oxide
* Presence of any medical or psychosocial condition, which the investigator believes, would hinder adherence to the study requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-28 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Emergent and Adverse Events | Baseline (day of kidney transplant surgery); 3, 14, 30, 90, 180, 270, and 365 days after starting study drug or placebo
  The difference in the proportion of cumulative treatment-emergent (TE) adverse events (AE) determined to be ≥ grade 3 severity that occur during 12 months from the first dose of FTY720 compared to the placebo group.

SECONDARY OUTCOMES:
Fraction of Renal Cortical Volume Occupied by Interstitium | Baseline, 3 months after kidney transplant, 1 year after kidney transplant
  A doubling of the fraction of renal cortical volume occupied by interstitium (VvInt/cortex) compared to the baseline biopsy in participants taking 0.5mg/day fingolimod (experimental group) or placebo (control group) for 3 months
MCP1 Biomarker | Baseline, 90 days, and 1 year after the first dose of fingolimod or placebo
  Measurement of Monocyte Chemoattractant Protein-1
Procollagen 3 Peptide Biomarker | Baseline, 90 days, and 1 year after the first dose of fingolimod or placebo
  Measurement of Procollagen 3 Peptide
BMP-7 Protein Biomarker | Baseline, 90 days, and 1 year after the first dose of fingolimod or placebo
  Measurement of Bone Morphogenetic Protein 7
TGF-beta Biomarker | Baseline, 90 days, and 1 year after the first dose of fingolimod or placebo
  Measurement of Transforming Growth Factor beta
RhoA of Blood Monocytes | Baseline, 90 days, and 1 year after the first dose of fingolimod or placebo
  Measurement of Ras homolog family member A protein
RICTOR Biomarker | Baseline, 90 days, and 1 year after the first dose of fingolimod or placebo
  Measurement of RPTOR Independent Companion Of MTOR Complex 2
Urinary Albumin:Creatinine Ratio | Baseline; 3, 14, 30, 90, 180, 270, and 365 days after starting study drug or placebo
  The ratio of albumin to creatinine in a urine sample from the patient
Change in Estimated Glomerular Filtration Rate | Baseline; 3, 14, 30, 90, 180, 270, and 365 days after starting study drug or placebo
  Estimated glomerular filtration rate relative to the baseline value or previous endpoints
Causes of End-Stage Renal Disease | Up to 1 year after taking the first dose of the study drug or placebo
  Recording the cause of end-stage renal disease, if it develops
Biopsy-Proven Acute Rejection | Baseline, 3 months after kidney transplant, 1 year after kidney transplant
  Biopsy-proven acute rejection as diagnosed by a qualified pathologist
Patient Survival | Baseline; 3, 14, 30, 90, 180, 270, and 365 days after starting study drug or placebo
  Whether the patient is deceased or alive
Graft Survival | Baseline; 3, 14, 30, 90, 180, 270, and 365 days after starting study drug or placebo
  Whether the patient required a new kidney graft or the patient is deceased

CONTACTS AND LOCATIONS:
Locations (1):
- Houston Methodist Research Institute, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gilenya [package insert]. East Hanover, NJ: Novartis Pharmaceuticals Corporation; 2019.
- [Background] Chen W, Chen W, Li XC, Ghobrial RM, Kloc M. Coinhibition of mTORC1/mTORC2 and RhoA/ROCK pathways prevents chronic rejection of rat cardiac allografts. Transplant Reports. 2018;3(4):21-28.
- [Background] Hart A, Smith JM, Skeans MA, Gustafson SK, Stewart DE, Cherikh WS, Wainright JL, Kucheryavaya A, Woodbury M, Snyder JJ, Kasiske BL, Israni AK. OPTN/SRTR 2015 Annual Data Report: Kidney. Am J Transplant. 2017 Jan;17 Suppl 1(Suppl 1):21-116. doi: 10.1111/ajt.14124. PMID 28052609
- [Background] Hart A, Smith JM, Skeans MA, Gustafson SK, Wilk AR, Castro S, Robinson A, Wainright JL, Snyder JJ, Kasiske BL, Israni AK. OPTN/SRTR 2017 Annual Data Report: Kidney. Am J Transplant. 2019 Feb;19 Suppl 2:19-123. doi: 10.1111/ajt.15274. PMID 30811893
- [Background] Matas AJ, Smith JM, Skeans MA, Thompson B, Gustafson SK, Stewart DE, Cherikh WS, Wainright JL, Boyle G, Snyder JJ, Israni AK, Kasiske BL. OPTN/SRTR 2013 Annual Data Report: kidney. Am J Transplant. 2015 Jan;15 Suppl 2:1-34. doi: 10.1111/ajt.13195. PMID 25626344
- [Background] OPTN/SRTR Annual Data Report - 2011. 2011; https://srtr.transplant.hrsa.gov/annual_reports/2011/Default.aspx. Accessed July 29, 2020.
- [Background] Vanhove T, Goldschmeding R, Kuypers D. Kidney Fibrosis: Origins and Interventions. Transplantation. 2017 Apr;101(4):713-726. doi: 10.1097/TP.0000000000001608. PMID 27941433
- [Background] Nankivell BJ, Chapman JR. Chronic allograft nephropathy: current concepts and future directions. Transplantation. 2006 Mar 15;81(5):643-54. doi: 10.1097/01.tp.0000190423.82154.01. PMID 16534463
- [Background] Meng XM, Nikolic-Paterson DJ, Lan HY. Inflammatory processes in renal fibrosis. Nat Rev Nephrol. 2014 Sep;10(9):493-503. doi: 10.1038/nrneph.2014.114. Epub 2014 Jul 1. PMID 24981817
- [Background] Sis B, Einecke G, Chang J, Hidalgo LG, Mengel M, Kaplan B, Halloran PF. Cluster analysis of lesions in nonselected kidney transplant biopsies: microcirculation changes, tubulointerstitial inflammation and scarring. Am J Transplant. 2010 Feb;10(2):421-30. doi: 10.1111/j.1600-6143.2009.02938.x. Epub 2010 Jan 6. PMID 20055794
- [Background] Naesens M, Kuypers DR, De Vusser K, Vanrenterghem Y, Evenepoel P, Claes K, Bammens B, Meijers B, Lerut E. Chronic histological damage in early indication biopsies is an independent risk factor for late renal allograft failure. Am J Transplant. 2013 Jan;13(1):86-99. doi: 10.1111/j.1600-6143.2012.04304.x. Epub 2012 Nov 8. PMID 23136888
- [Background] Nankivell BJ, Fenton-Lee CA, Kuypers DR, Cheung E, Allen RD, O'Connell PJ, Chapman JR. Effect of histological damage on long-term kidney transplant outcome. Transplantation. 2001 Feb 27;71(4):515-23. doi: 10.1097/00007890-200102270-00006. PMID 11258430
- [Background] Cosio FG, Grande JP, Larson TS, Gloor JM, Velosa JA, Textor SC, Griffin MD, Stegall MD. Kidney allograft fibrosis and atrophy early after living donor transplantation. Am J Transplant. 2005 May;5(5):1130-6. doi: 10.1111/j.1600-6143.2005.00811.x. PMID 15816896
- [Background] Nankivell BJ, Borrows RJ, Fung CL, O'Connell PJ, Allen RD, Chapman JR. The natural history of chronic allograft nephropathy. N Engl J Med. 2003 Dec 11;349(24):2326-33. doi: 10.1056/NEJMoa020009. PMID 14668458
- [Background] Fioretto P, Steffes MW, Sutherland DE, Mauer M. Sequential renal biopsies in insulin-dependent diabetic patients: structural factors associated with clinical progression. Kidney Int. 1995 Dec;48(6):1929-35. doi: 10.1038/ki.1995.493. PMID 8587254
- [Background] Ibrahim HN, Jackson S, Connaire J, Matas A, Ney A, Najafian B, West A, Lentsch N, Ericksen J, Bodner J, Kasiske B, Mauer M. Angiotensin II blockade in kidney transplant recipients. J Am Soc Nephrol. 2013 Feb;24(2):320-7. doi: 10.1681/ASN.2012080777. Epub 2013 Jan 10. PMID 23308016
- [Background] Budde K, Schmouder RL, Brunkhorst R, Nashan B, Lucker PW, Mayer T, Choudhury S, Skerjanec A, Kraus G, Neumayer HH. First human trial of FTY720, a novel immunomodulator, in stable renal transplant patients. J Am Soc Nephrol. 2002 Apr;13(4):1073-1083. doi: 10.1681/ASN.V1341073. PMID 11912269
- [Background] Kovarik JM, Schmouder R, Barilla D, Wang Y, Kraus G. Single-dose FTY720 pharmacokinetics, food effect, and pharmacological responses in healthy subjects. Br J Clin Pharmacol. 2004 May;57(5):586-91. doi: 10.1111/j.1365-2125.2003.02065.x. PMID 15089811
- [Background] Kovarik JM, Schmouder R, Barilla D, Riviere GJ, Wang Y, Hunt T. Multiple-dose FTY720: tolerability, pharmacokinetics, and lymphocyte responses in healthy subjects. J Clin Pharmacol. 2004 May;44(5):532-7. doi: 10.1177/0091270004264165. PMID 15102874
- [Background] Bohler T, Waiser J, Schuetz M, Neumayer HH, Budde K. FTY720 exerts differential effects on CD4+ and CD8+ T-lymphocyte subpopulations expressing chemokine and adhesion receptors. Nephrol Dial Transplant. 2004 Mar;19(3):702-13. doi: 10.1093/ndt/gfg599. PMID 14767029
- [Background] Kahan BD, Karlix JL, Ferguson RM, Leichtman AB, Mulgaonkar S, Gonwa TA, Skerjanec A, Schmouder RL, Chodoff L. Pharmacodynamics, pharmacokinetics, and safety of multiple doses of FTY720 in stable renal transplant patients: a multicenter, randomized, placebo-controlled, phase I study. Transplantation. 2003 Oct 15;76(7):1079-84. doi: 10.1097/01.TP.0000084822.01372.AC. PMID 14557756
- [Background] Park SI, Felipe CR, Machado PG, Garcia R, Skerjanec A, Schmouder R, Tedesco-Silva H Jr, Medina-Pestana JO. Pharmacokinetic/pharmacodynamic relationships of FTY720 in kidney transplant recipients. Braz J Med Biol Res. 2005 May;38(5):683-94. doi: 10.1590/S0100-879X2005000500005. Epub 2005 May 25. PMID 15917949
- [Background] Skerjanec A, Tedesco H, Neumayer HH, Cole E, Budde K, Hsu CH, Schmouder R. FTY720, a novel immunomodulator in de novo kidney transplant patients: pharmacokinetics and exposure-response relationship. J Clin Pharmacol. 2005 Nov;45(11):1268-78. doi: 10.1177/0091270005279799. PMID 16239360
- [Background] Mulgaonkar S, Tedesco H, Oppenheimer F, Walker R, Kunzendorf U, Russ G, Knoflach A, Patel Y, Ferguson R; FTYA121 study group. FTY720/cyclosporine regimens in de novo renal transplantation: a 1-year dose-finding study. Am J Transplant. 2006 Aug;6(8):1848-57. doi: 10.1111/j.1600-6143.2006.01404.x. Epub 2006 Jun 12. PMID 16771816
- [Background] Salvadori M, Budde K, Charpentier B, Klempnauer J, Nashan B, Pallardo LM, Eris J, Schena FP, Eisenberger U, Rostaing L, Hmissi A, Aradhye S; FTY720 0124 Study Group. FTY720 versus MMF with cyclosporine in de novo renal transplantation: a 1-year, randomized controlled trial in Europe and Australasia. Am J Transplant. 2006 Dec;6(12):2912-21. doi: 10.1111/j.1600-6143.2006.01552.x. PMID 17061999
- [Background] Tedesco-Silva H, Szakaly P, Shoker A, Sommerer C, Yoshimura N, Schena FP, Cremer M, Hmissi A, Mayer H, Lang P; FTY720 2218 Clinical Study Group. FTY720 versus mycophenolate mofetil in de novo renal transplantation: six-month results of a double-blind study. Transplantation. 2007 Oct 15;84(7):885-92. doi: 10.1097/01.tp.0000281385.26500.3b. PMID 17984842
- [Background] Tedesco-Silva H, Lorber MI, Foster CE, Sollinger HW, Mendez R, Carvalho DB, Shapiro R, Rajagopalan PR, Mayer H, Slade J, Kahan BD; FTY720A2202 clinical study group. FTY720 and everolimus in de novo renal transplant patients at risk for delayed graft function: results of an exploratory one-yr multicenter study. Clin Transplant. 2009 Sep-Oct;23(5):589-99. doi: 10.1111/j.1399-0012.2009.01070.x. Epub 2009 Aug 27. PMID 19719728
- [Background] Hoitsma AJ, Woodle ES, Abramowicz D, Proot P, Vanrenterghem Y; FTY720 Phase II Transplant Study Group. FTY720 combined with tacrolimus in de novo renal transplantation: 1-year, multicenter, open-label randomized study. Nephrol Dial Transplant. 2011 Nov;26(11):3802-5. doi: 10.1093/ndt/gfr503. Epub 2011 Sep 12. PMID 21911597
- [Background] Kappos L, Antel J, Comi G, Montalban X, O'Connor P, Polman CH, Haas T, Korn AA, Karlsson G, Radue EW; FTY720 D2201 Study Group. Oral fingolimod (FTY720) for relapsing multiple sclerosis. N Engl J Med. 2006 Sep 14;355(11):1124-40. doi: 10.1056/NEJMoa052643. PMID 16971719
- [Background] Chen W, Chen S, Chen W, Li XC, Ghobrial RM, Kloc M. Screening RhoA/ROCK inhibitors for the ability to prevent chronic rejection of mouse cardiac allografts. Transpl Immunol. 2018 Oct;50:15-25. doi: 10.1016/j.trim.2018.06.002. Epub 2018 Jun 6. PMID 29885441
- [Background] Chen W, Ghobrial RM, Li XC, Kloc M. Inhibition of RhoA and mTORC2/Rictor by Fingolimod (FTY720) induces p21-activated kinase 1, PAK-1 and amplifies podosomes in mouse peritoneal macrophages. Immunobiology. 2018 Nov;223(11):634-647. doi: 10.1016/j.imbio.2018.07.009. Epub 2018 Jul 7. PMID 30005970
- [Background] CONSORT Group. CONSORT Transparent reporting of trials. 2010; http://www.consort-statement.org/consort-2010. Accessed July 29, 2020.
- [Background] Budde K, L Schmouder R, Nashan B, Brunkhorst R, W Lucker P, Mayer T, Brookman L, Nedelman J, Skerjanec A, Bohler T, Neumayer HH. Pharmacodynamics of single doses of the novel immunosuppressant FTY720 in stable renal transplant patients. Am J Transplant. 2003 Jul;3(7):846-54. doi: 10.1034/j.1600-6143.2003.00130.x. PMID 12814476